CLINICAL TRIAL: NCT05240872
Title: Is There Any Advantage of PRP Over Autologous Blood Injection in the Treatment of Chronic Plantar Fasciitis? A Prospective Randomized Double Blinded Study
Brief Title: Effects of Autologous Blood Injection Versus Platelet Rich Plasma on Chronic Plantar Fasciitis
Acronym: PF:AutovsPRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ozcan Kaya, Orthopaedics and Traumatology Specialist, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13.02.2020/008
Record Dates: First submitted 2022-02-13; First posted 2022-02-15 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Plantar Fascitis
Keywords: heel pain, platelet rich plasm, autologous blood injection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Platelet Rich Plasm (PRP) injection group
  Interventions: Biological: PRP injection
- Group B (Active Comparator): Autologous Blood injection (ABI) group
  Interventions: Biological: ABI injection

INTERVENTIONS:
Biological: PRP injection — Plantar fascia injection therapy with PRP
  Arms: Group A
Biological: ABI injection — ABI injection
  Arms: Group B

SUMMARY:
To explore effects of Autologous Blood Injection versus Platelet Rich plasma injection for treatment of chronic plantar fasciitis

DETAILED DESCRIPTION:
After clinical diagnosis of patients with plantar fasciitis. Patients were divided into two groups. Group A (PRP injection group) and Group B (ABI group) were randomized according to web based block group randomization. Patients were evaluated prior to injection in terms of Health related quality of life scores related to foot and ankle diseases (AOFAS and FADI) and VAS. After injection at 1st, 3rd and 6th months HRQoL were compared between groups. Intra group evaluation for HRQoL were performed at f/up visits. Independent t test and repeated measure ANOVA test used for statistical analysis

ELIGIBILITY:
Inclusion Criteria:

1. Participants who were diagnosed with chronic plantar fasciitis
2. Nonresponded to o conservative treatment (stretching exercises, nonsteroidal anti-inflammatory drugs, and heel pads) for at least 6 weeks
3. Patient should be able to understand the informed consent about type of treatment and blindness and randomization
4. Visual analog scale pain higher than 5 (on a 10-point visual analog scale)

Exclusion Criteria:

1. previous history of any type of local injection treatment for heel pain
2. history of surgery for heel pain, foot and ankle disorders, fractures
3. Associated pathology involving the lower limb such as

   * tarsal tunnel syndrome
   * effusion of the ankle indicating an intra-articular disease
   * Peroneal/Achilles/tibialis tendons pathology
   * any obvious deformity of foot and ankle,
4. Patients with systemic disorder like diabetes mellitus, ankylosing spondylitis rheumatoid arthritis, hematological disease, or gout
5. Pregnancy
6. Use of antiocoagulation -

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Changes in Visual Analogue Scale (VAS) | 0,1 st 3rd and 6th month; changes between time points will be assessed
  Visual Analogue Scale 10 worst 0-1 best in terms of pain outcome
Changes in American Orthopaedic Foot & Ankle Society (AOFAS ) Score | 0,1 st 3rd and 6th month; changes between time points will be assessed
  American Orthopaedic Foot & Ankle Society (AOFAS) Clinical rating systems for the ankle-hindfoot, midfoot, hallux, and lesser toes Evaluation:0 worst 100 best
Changes in Foot and Ankle Disability Index (FADI) | 0,1 st 3rd and 6th month; changes between time points will be assessed
  Foot and Ankle Disability Index Evaluation:0 worst 100 best

CONTACTS AND LOCATIONS:
Overall Officials: Celalettin Bildik, MD, Principal Investigator — Istanbul Atasehir Florence Nightingale Hospital
Locations (1):
- Atasehir Florence Nightingale Hospital, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
According to permission of Institutional Review of Board and Ethical Committee; Participating demographics, outcome measures may be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After acceptance to publish
Access Criteria: permission of Institutional Review of Board and Ethical Committee

REFERENCES:
- [Background] Kalia RB, Singh V, Chowdhury N, Jain A, Singh SK, Das L. Role of Platelet Rich Plasma in Chronic Plantar Fasciitis: A Prospective Study. Indian J Orthop. 2020 Oct 6;55(Suppl 1):142-148. doi: 10.1007/s43465-020-00261-w. eCollection 2021 May. PMID 34122767
- [Background] Latt LD, Jaffe DE, Tang Y, Taljanovic MS. Evaluation and Treatment of Chronic Plantar Fasciitis. Foot Ankle Orthop. 2020 Feb 13;5(1):2473011419896763. doi: 10.1177/2473011419896763. eCollection 2020 Jan. PMID 35097359
- [Background] Bagcier F, Yilmaz N. The Impact of Extracorporeal Shock Wave Therapy and Dry Needling Combination on Pain and Functionality in the Patients Diagnosed with Plantar Fasciitis. J Foot Ankle Surg. 2020 Jul-Aug;59(4):689-693. doi: 10.1053/j.jfas.2019.09.038. Epub 2020 Apr 25. PMID 32340838
- [Background] Landorf KB. Plantar heel pain and plantar fasciitis. BMJ Clin Evid. 2015 Nov 25;2015:1111. PMID 26609884
- [Background] Stuber K, Kristmanson K. Conservative therapy for plantar fasciitis: a narrative review of randomized controlled trials. J Can Chiropr Assoc. 2006 Jun;50(2):118-33. PMID 17549177
- [Background] Martin JE, Hosch JC, Goforth WP, Murff RT, Lynch DM, Odom RD. Mechanical treatment of plantar fasciitis. A prospective study. J Am Podiatr Med Assoc. 2001 Feb;91(2):55-62. doi: 10.7547/87507315-91-2-55. PMID 11266478
- [Background] Kaya O, Hurel C, Gumussuyu G, Kose O. Bilateral calcaneal insufficiency fractures due to chronic carbamazepine use for trigeminal neuralgia: A case report. Niger J Clin Pract. 2020 Apr;23(4):574-576. doi: 10.4103/njcp.njcp_515_18. PMID 32246668
- [Background] Gupta R, Malhotra A, Masih GD, Khanna T, Kaur H, Gupta P, Kashyap S. Comparing the Role of Different Treatment Modalities for Plantar Fasciitis: A Double Blind Randomized Controlled Trial. Indian J Orthop. 2020 Jan 20;54(1):31-37. doi: 10.1007/s43465-019-00038-w. eCollection 2020 Feb. PMID 32257015
- [Background] Mahindra P, Yamin M, Selhi HS, Singla S, Soni A. Chronic Plantar Fasciitis: Effect of Platelet-Rich Plasma, Corticosteroid, and Placebo. Orthopedics. 2016 Mar-Apr;39(2):e285-9. doi: 10.3928/01477447-20160222-01. Epub 2016 Feb 25. PMID 26913766
- [Background] Singh P, Madanipour S, Bhamra JS, Gill I. A systematic review and meta-analysis of platelet-rich plasma versus corticosteroid injections for plantar fasciopathy. Int Orthop. 2017 Jun;41(6):1169-1181. doi: 10.1007/s00264-017-3470-x. Epub 2017 Apr 10. PMID 28396927
- [Background] Jain SK, Suprashant K, Kumar S, Yadav A, Kearns SR. Comparison of Plantar Fasciitis Injected With Platelet-Rich Plasma vs Corticosteroids. Foot Ankle Int. 2018 Jul;39(7):780-786. doi: 10.1177/1071100718762406. Epub 2018 Mar 30. PMID 29600719
- [Background] Yu T, Xia J, Li B, Zhou H, Yang Y, Yu G. Outcomes of platelet-rich plasma for plantar fasciopathy: a best-evidence synthesis. J Orthop Surg Res. 2020 Sep 21;15(1):432. doi: 10.1186/s13018-020-01783-7. PMID 32958046
- [Background] Thomas JL, Christensen JC, Kravitz SR, Mendicino RW, Schuberth JM, Vanore JV, Weil LS Sr, Zlotoff HJ, Bouche R, Baker J; American College of Foot and Ankle Surgeons heel pain committee. The diagnosis and treatment of heel pain: a clinical practice guideline-revision 2010. J Foot Ankle Surg. 2010 May-Jun;49(3 Suppl):S1-19. doi: 10.1053/j.jfas.2010.01.001. PMID 20439021
- [Background] Shetty SH, Dhond A, Arora M, Deore S. Platelet-Rich Plasma Has Better Long-Term Results Than Corticosteroids or Placebo for Chronic Plantar Fasciitis: Randomized Control Trial. J Foot Ankle Surg. 2019 Jan;58(1):42-46. doi: 10.1053/j.jfas.2018.07.006. Epub 2018 Nov 15. PMID 30448183
- [Background] Crawford F, Atkins D, Young P, Edwards J. Steroid injection for heel pain: evidence of short-term effectiveness. A randomized controlled trial. Rheumatology (Oxford). 1999 Oct;38(10):974-7. doi: 10.1093/rheumatology/38.10.974. PMID 10534548
- [Background] Tsai WC, Hsu CC, Chen CP, Chen MJ, Yu TY, Chen YJ. Plantar fasciitis treated with local steroid injection: comparison between sonographic and palpation guidance. J Clin Ultrasound. 2006 Jan;34(1):12-6. doi: 10.1002/jcu.20177. PMID 16353228
- [Background] Tatli YZ, Kapasi S. The real risks of steroid injection for plantar fasciitis, with a review of conservative therapies. Curr Rev Musculoskelet Med. 2009 Mar;2(1):3-9. doi: 10.1007/s12178-008-9036-1. Epub 2008 Sep 19. PMID 19468912
- [Background] Arnoczky SP, Sheibani-Rad S. The basic science of platelet-rich plasma (PRP): what clinicians need to know. Sports Med Arthrosc Rev. 2013 Dec;21(4):180-5. doi: 10.1097/JSA.0b013e3182999712. PMID 24212364
- [Background] Foster TE, Puskas BL, Mandelbaum BR, Gerhardt MB, Rodeo SA. Platelet-rich plasma: from basic science to clinical applications. Am J Sports Med. 2009 Nov;37(11):2259-72. doi: 10.1177/0363546509349921. PMID 19875361
- [Background] Hall MP, Band PA, Meislin RJ, Jazrawi LM, Cardone DA. Platelet-rich plasma: current concepts and application in sports medicine. J Am Acad Orthop Surg. 2009 Oct;17(10):602-8. doi: 10.5435/00124635-200910000-00002. PMID 19794217
- [Background] Ragab EM, Othman AM. Platelets rich plasma for treatment of chronic plantar fasciitis. Arch Orthop Trauma Surg. 2012 Aug;132(8):1065-70. doi: 10.1007/s00402-012-1505-8. Epub 2012 May 4. PMID 22555761
- [Background] Martinelli N, Marinozzi A, Carni S, Trovato U, Bianchi A, Denaro V. Platelet-rich plasma injections for chronic plantar fasciitis. Int Orthop. 2013 May;37(5):839-42. doi: 10.1007/s00264-012-1741-0. Epub 2012 Dec 19. PMID 23250352
- [Background] Wheeler PC, Dudson C. Similar Benefits Seen After Radial Extracorporeal Shockwave Therapy or Autologous Blood Injection in Patients With Chronic Plantar Fasciitis-A Retrospective Cohort Study. Clin J Sport Med. 2022 Mar 1;32(2):e107-e115. doi: 10.1097/JSM.0000000000000930. PMID 34267064
- [Background] Lee TG, Ahmad TS. Intralesional autologous blood injection compared to corticosteroid injection for treatment of chronic plantar fasciitis. A prospective, randomized, controlled trial. Foot Ankle Int. 2007 Sep;28(9):984-90. doi: 10.3113/FAI.2007.0984. PMID 17880872
- [Background] Karimzadeh A, Raeissadat SA, Erfani Fam S, Sedighipour L, Babaei-Ghazani A. Autologous whole blood versus corticosteroid local injection in treatment of plantar fasciitis: A randomized, controlled multicenter clinical trial. Clin Rheumatol. 2017 Mar;36(3):661-669. doi: 10.1007/s10067-016-3484-6. Epub 2016 Dec 12. PMID 27957618
- [Background] Tsikopoulos K, Tsikopoulos A, Natsis K. Autologous whole blood or corticosteroid injections for the treatment of epicondylopathy and plantar fasciopathy? A systematic review and meta-analysis of randomized controlled trials. Phys Ther Sport. 2016 Nov;22:114-122. doi: 10.1016/j.ptsp.2016.02.002. Epub 2016 Feb 24. PMID 27085490